CLINICAL TRIAL: NCT03407963
Title: Feasibility of Prostatic Arterial Embolization in Low-risk Patients With Unilateral Prostate Cancer Under Active Surveillance: Monocentric Pilot Study
Acronym: CAPEMBOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIMAO/2017-01/JF-01; 2017-A01915-48 (Other: ANSM)
Record Dates: First submitted 2018-01-09; First posted 2018-01-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Embolization, Therapeutic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate cancer patients (Experimental)
  Interventions: Procedure: Embolization

INTERVENTIONS:
Procedure: Embolization — Embolization by microparticles (300-500 microns)

SUMMARY:
The authors hypothesize that, in patients with low volume tumors identified according to anatomo-pathological criteria and imaging, and under active surveillance focal, therapy by unilateral embolization of prostatic arteries will provide local control of the tumor via selective ischemia

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is between 18 and 80 years old
* Patient has unilateral prostate cancer, stage TNM<T2b with an MRI PiRAds target ≥ 3 in concordance with biopsy result
* Biopsy gives a Gleason score ≤ 6 with more than 3 positive biopsies per lob and at least 50% the length of the positive biopsy; patients over 70 years old with a Gleason score = 7 (3+4) can be included
* Patient has a life expectancy of over 10 years
* PSA <10ng/ml; patients with a large prostatic volume and PSA ≥ 10ng/ml can be included according to doctor discretion.

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient unresponsive to active surveillance
* Patient refusing active surveillance
* Patients in a state unfit to express personal consent cannot be solicited (eg patients undergoing psychiatric treatment with mental difficulties rendering consent impossible)
* Contraindication for MRI (pacemaker incompatible with MRI, claustrophobia, metal device, prosthetic hip replacement)
* Patient with hemostasis disorder.
* Cancer in both prostate lobes

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Complications arising from embolization | Month 6
  Presence/absence of complications beyond those expected linked to embolization (persistent urinary infection, dysuria, rectorrhagia, hematuria, hemospermia, acute urinary retention and pelvic perineal pain)
Presence of cancerous cells | Month 6
  Positive/negative according to biopsy of treated lobe

SECONDARY OUTCOMES:
Global survival | Month 6
  days
Use of other mode of treatment | Month 1
  Yes/No of radical treatment (surgery, radiotherapy, high intensity focused ultrasound)
Use of other mode of treatment | Month 3
  Yes/No of radical treatment (surgery, radiotherapy, high intensity focused ultrasound)
Use of other mode of treatment | Month 6
  Yes/No of radical treatment (surgery, radiotherapy, high intensity focused ultrasound)
Necrosis of treated lobe | Day 0
  MRI analysis (Pi RADS VS and RECIST 1.1 if lesion >10mm)
Necrosis of treated lobe | Week 2
  MRI analysis (Pi RADS VS and RECIST 1.1 if lesion >10mm)
Necrosis of treated lobe | Month 6
  MRI analysis (Pi RADS VS and RECIST 1.1 if lesion >10mm)
Change in size of target | Day 0
  MRI analysis (Pi RADS VS and RECIST 1.1 if lesion >10mm)
Change in size of target | Week 2
  MRI analysis (Pi RADS VS and RECIST 1.1 if lesion >10mm)
Change in size of target | Month 6
  MRI analysis (Pi RADS VS and RECIST 1.1 if lesion >10mm)
Prostate specific antigen level | Month 1
  ng/ml
Prostate specific antigen level | Month 3
  ng/ml
Prostate specific antigen level | Month 6
  ng/ml
Occurrence of undesirable events linked to embolization or the femoral access classified according to Clavien-Dindo classification | Month 1
  Expected events: severe allergic reaction to contrast product, septicemia with urinary origin, persistent urinary infection, dysuria, serious hematuria, hemospermia, bladder ulceration/necrosis, rectal ulcer, rectorrhagia, irradiation-induced severe epidermal lesions, acute urinary retention, pelvic-perineal pain, prostatitis, epididymitis, obstructive renal failure, chronic bladder retention, lithiasis, hypocontractile bladder, elevation of PSA (at 6 months linked to probable disease progression).
Occurrence of undesirable events linked to embolization or the femoral access classified according to Clavien-Dindo classification | Month 3
  Expected events: severe allergic reaction to contrast product, septicemia with urinary origin, persistent urinary infection, dysuria, serious hematuria, hemospermia, bladder ulceration/necrosis, rectal ulcer, rectorrhagia, irradiation-induced severe epidermal lesions, acute urinary retention, pelvic-perineal pain, prostatitis, epididymitis, obstructive renal failure, chronic bladder retention, lithiasis, hypocontractile bladder, elevation of PSA (at 6 months linked to probable disease progression).
Occurrence of undesirable events linked to embolization or the femoral access classified according to Clavien-Dindo classification | Month 6
  Expected events: severe allergic reaction to contrast product, septicemia with urinary origin, persistent urinary infection, dysuria, serious hematuria, hemospermia, bladder ulceration/necrosis, rectal ulcer, rectorrhagia, irradiation-induced severe epidermal lesions, acute urinary retention, pelvic-perineal pain, prostatitis, epididymitis, obstructive renal failure, chronic bladder retention, lithiasis, hypocontractile bladder, elevation of PSA (at 6 months linked to probable disease progression).
Urinary symptoms | Month 1
  International Prostate Symptom Score (IPSS score) (0-35)
Urinary symptoms | Month 3
  International Prostate Symptom Score (IPSS score) (0-35)
Urinary symptoms | Month 6
  International Prostate Symptom Score (IPSS score) (0-35)
Incontinence | Month 1
  24-hr pad test (g)
Incontinence | Month 3
  24-hr pad test (g)
Incontinence | Month 6
  24-hr pad test (g)
Erectile dysfunction | Month 1
  International Index of Erectile Function (IIEF-6) questionnaire (score 0-30)
Erectile dysfunction | Month 3
  International Index of Erectile Function (IIEF-6) questionnaire (score 0-30)
Erectile dysfunction | Month 6
  International Index of Erectile Function (IIEF-6) questionnaire (score 0-30)
Health-related quality of life | Month 1
  euroqol 5 dimension questionnaire (EQ-5D)
Health-related quality of life | Month 3
  euroqol 5 dimension questionnaire (EQ-5D)
Health-related quality of life | Month 6
  euroqol 5 dimension questionnaire (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Frandon, MD, Study Director — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Result] Frandon J, Bey E, Hamard A, Mohammad H, Gonzalez S, Greffier J, Chevallier T, de Forges H, Beregi JP, Droupy S. Early Results of Unilateral Prostatic Artery Embolization as a Focal Therapy in Patients with Prostate Cancer under Active Surveillance: Cancer Prostate Embolisation, a Pilot Study. J Vasc Interv Radiol. 2021 Feb;32(2):247-255. doi: 10.1016/j.jvir.2020.10.002. Epub 2020 Nov 25. PMID 33248919